CLINICAL TRIAL: NCT04939610
Title: LuMIERE: A Phase 1/2, Multicenter, Open-label, Non-randomized Study to Investigate Safety and Tolerability, Pharmacokinetics, Dosimetry, and Preliminary Activity of 177Lu-FAP-2286 in Patients With an Advanced Solid Tumor
Brief Title: A Study of 177Lu-FAP-2286 in Advanced Solid Tumors
Acronym: LuMIERE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CO-2286-114; CAAA614A12101 (Other: Novartis); 2023-508995-12-00 (Other: EU CTIS registry)
Record Dates: First submitted 2021-06-09; First posted 2021-06-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor
Keywords: 177Lu-FAP-2286; 68Ga-FAP-2286; Theranostic; FAP-2286; Fibroblast Activation Protein (FAP); Dosimetry; cancer-associated fibroblasts (CAF); Peptide-Targeted Radioligand Therapy (PTRT); Peptide Receptor Radionuclide Therapy (PRRT); Targeted radioligand therapy (TRT); Targeted radionuclide therapy; Lutetium-177; Gallium-68

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose Escalation (Experimental): Up to 30 patients with solid tumors.
  Interventions: Drug: 68Ga-FAP-2286; Drug: 177Lu-FAP-2286
- Phase 2: Specific Solid Tumors (Experimental): Up to 192 participants treated with [177Lu]Lu-FAP-2286 in tumor-specific participant groups in monotherapy and in combination with chemotherapy.
  Interventions: Drug: 68Ga-FAP-2286; Drug: 177Lu-FAP-2286

INTERVENTIONS:
Drug: 68Ga-FAP-2286 — 68Ga-FAP-2286 IV administered as imaging agent for PET scan.
Drug: 177Lu-FAP-2286 — Phase 1:
  Patients with positive uptake of 68Ga-FAP- 2286 will receive a fixed dose of 177Lu-FAP-2286 IV administered every 6 weeks for a maximum of 6 doses. Doses range between 3.7 and 9.25 GBq (100-250 mCi).
  Phase 2:
  Monotherapy: Patients with positive uptake of 68Ga FAP 2286 will receive a fixed dose of 177Lu FAP 2286 IV administered at the RP2D determined in Phase 1 dose escalation in every 4 weeks.
  Combination therapy: Patients with positive uptake of 68Ga FAP 2286 will receive 177Lu-FAP-2286 based on dose escalation (starting with dose level 1) followed by dose expansion at selected dose.

SUMMARY:
Fibroblast activation protein (FAP) is a cell surface protein that is highly expressed on the surface of cancer-associated fibroblasts (CAFs) present in the tumor microenvironment of most epithelial cancers, whereas limited expression of FAP is observed in normal tissues. In some cancers of mesenchymal origin, notably sarcoma and mesothelioma, FAP expression has also been observed on the tumor cells themselves. Given the restricted expression profile, FAP is a promising target for peptide-targeted radionuclide imaging and therapeutic agents.

Phase 1 of this study is designed to evaluate the safety and establish the recommended intravenous (IV) Phase 2 dose (RP2D) for [177Lu]Lu FAP 2286 monotherapy in participants with FAP expressing solid tumors.

Phase 2 is designed to evaluate the safety and efficacy of [177Lu]Lu FAP 2286 as monotherapy in participants with pancreatic ductal adenocarcinoma (PDAC), non-small cell lung cancer (NSCLC), and breast cancer (BC) and in combination with chemotherapy in participants with untreated PDAC or relapsed NSCLC.

Participants in both Phase 1 and 2 will be selected for treatment with [177Lu]Lu FAP 2286 based on [68Ga]Ga FAP 2286 imaging for determining tumor FAP expression.

DETAILED DESCRIPTION:
Screening Period:

All participants will undergo screening assessments including disease assessments per CT or MRI per RECIST v1.1 criteria prior to administration of [68Ga]Ga FAP 2286. Each participant must provide informed consent and agree to provide an archival tumor tissue sample, if available, and blood samples for biomarker assessment. Participants must meet all entry criteria as specified in the protocol.

In Phase 1 only, participants will also undergo FDG-PET imaging. In the Phase 2 part, [177Lu]Lu FAP 2286 will be investigated in monotherapy and in combination with chemotherapy. All participants in the combination group may begin chemotherapy prior to [177Lu]Lu FAP 2286.

Participants meeting entry criteria will be enrolled and participants who have not had prior PET/CT imaging with [68Ga]Ga FAP 2286 in the previous 3 months (applicable only to Phase 1) will undergo PET imaging with [68Ga]Ga FAP prior to initiating treatment with [177Lu]Lu FAP 2286. Participants must have a positive [68Ga]Ga FAP PET/CT scan, as described in the criteria for continuation to [177Lu]Lu FAP 2286 therapy, in order to be treated with [177Lu]Lu FAP 2286.

Treatment Period:

A single IV dose of [177Lu]Lu FAP 2286 will be initially administered every 6 weeks (window of - 1 to + 7 days) up to a maximum of 6 doses in Phase 1. In Phase 2, [177Lu]Lu FAP 2286 will be administered every 4 weeks (28 days ± 3 days).

All participants will be monitored for safety throughout the Treatment Period. All participants will be assessed for disease status per RECIST v1.1 every 6 weeks (42 days). Participants will receive [177Lu]Lu FAP 2286 until the maximum doses allowed are administered, confirmed radiographic disease progression assessed by investigator based on RECIST v1.1 criteria, unequivocal clinical disease progression, unacceptable toxicity or inability to tolerate further treatment, loss to follow-up, or withdrawal of consent.

Safety data will be periodically reviewed by the DCRC during dose escalation and by a Data Monitoring Committee (DMC) during dose expansion.

End of Treatment (EOT) Visit:

In Phase 1, participants will have an EOT Visit 6 to 8 weeks after the last dose of [177Lu]Lu FAP 2286 except in cases of participant death, loss to follow up, or withdrawal of consent for further follow up. Participants in Phase 2 will have an EOT visit within 28 days from the last dose of study treatment except in case of participant death, loss to follow-up, or withdrawal of consent for further follow-up.

Post treatment safety follow-up:

In Phase 2, after discontinuation of study treatment for any reason, all participants will have safety follow-up for 6 weeks (+/- 1 week) after their last study treatment administration, except in case of death, loss to follow-up or withdrawal of consent as per the schedule of assessments.

Long-term Follow-up (LFTU) Period:

Upon completion of the EOT Visit, participants will enter the LTFU Period. The LTFU Period will include safety, disease, and survival assessments, as applicable.

* Safety assessments will be performed every 12 weeks (+/- 1 week) for 2 years, then every 6 months until 5 years.
* Disease assessments will be performed for all participants who complete the EOT for a reason other than radiographic disease progression. Participants should continue to have tumor scans performed until radiographic disease progression, death, loss to follow-up, withdrawal from study, study closure or initiation of subsequent anticancer treatment.
* Survival assessments will be performed for all participants.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must meet the following inclusion criteria. The criteria below apply to participants enrolling in Phase 1 and Phase 2, unless otherwise specified.

1. Have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved Informed Consent Form (ICF) prior to any study-specific evaluation.
2. Be ≥ 18 years of age at the time the ICF is signed.
3. Have consented to submission of fresh or archival tumor tissue, if available.
4. Have adequate organ function confirmed by the following laboratory values obtained within the Screening Period prior to administration of [68Ga]Ga FAP 2286 and prior to first cycle of chemotherapy in the combination groups:

   a. Bone Marrow Function (independent of transfusion or growth factor support within 21 days prior to planned first administration of [177Lu]Lu FAP 2286): i. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; ii. Platelets > 100 × 109/L; and iii.Hemoglobin ≥ 9 g/dL. b. Hepatic Function: i. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × institutional upper limit of normal (ULN); if liver metastases, then ≤ 5 × the institutional ULN; ii. Serum Bilirubin ≤ 1.5 × institutional ULN or if known Gilbert's syndrome then ≤ 3 × institutional ULN; iii. Serum albumin ≥ 30 g/L (3 g/dL) and iv. INR ≤ 1.5 x ULN and activated partial thromboplastin time (aPTT)≤1.5 x ULN. This applies to participants who are not receiving therapeutic anticoagulation, participants receiving therapeutic anticoagulation should be on a stable dose.

   c. Renal Function: i. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min using the Cockcroft Gault formula.
5. Have an Eastern Oncology Group (ECOG) performance status of 0 or 1.
6. Have a life expectancy of ≥ 6 months.
7. Have measurable disease per RECIST v1.1 meeting the following criteria:

   1. At least 1 lesion of ≥ 10 mm in the longest diameter for a non lymph node or ≥ 15 mm in the short axis diameter for a lymph node that is serially measurable according to RECIST v1.1 using conventional CT and/or MRI.

      • Lesions that have had external beam radiotherapy or loco-regional therapies such as radiofrequency ablation must show subsequent evidence of substantial size increase to be deemed a target lesion.

      For Phase 1 only:
8. Have a histologically and/or cytologically confirmed advanced/metastatic solid tumor not amenable to treatment with curative intent:

   a. Tumor must be refractory to or have progressed following prior treatment and have no satisfactory alternative treatment options.

   For Phase 2 only:
9. Have cytologically or histologically and radiologically confirmed recurrent or metastatic disease as outlined below:

   a. Pancreatic Cancer monotherapy group: i. Pancreatic ductal adenocarcinoma (ductal adenocarcinoma and related subtypes eligible; endocrine and neuroendocrine tumors excluded) ii. Participants must have progressed after at least 1, but no more than two prior chemotherapy regimens for locally advanced unresectable or metastatic disease.

   Criteria b through h removed during Protocol amendment 7. i. Pancreatic Cancer combination group (with mFOLFIRINOX) i. Pancreatic ductal adenocarcinoma (ductal adenocarcinoma and related subtypes eligible; endocrine and neuroendocrine tumors excluded); ii. Participants have not received prior systemic therapy for metastatic disease.

   j. Non-small cell lung cancer monotherapy group i. Non-small cell lung cancer (adenocarcinoma and squamous eligible; endocrine, neuroendocrine and small cell tumors are excluded) ii. Participants must have progressed after at least 1 but not more than 2 prior systemic regimens including chemotherapy and immunotherapy. Participants with NSCLC and targeted therapy treatment options, are eligible for the clinical trial as long as they meet these criteria (progression after 1 or 2 prior therapies). Note: Participants with NSCLC harboring mutations amenable to targeted therapy treatment, are eligible if received targeted therapy as single agent or in combination in 1st or 2nd line of treatment; participants not eligible to receive such therapies in 1st or 2nd line are also eligible to participate to the study.

   iii. Participants who have received adjuvant or neoadjuvant platinum-doublet chemotherapy (after surgery and/or radiation therapy) and an immune checkpoint inhibitor and developed recurrent or metastatic disease while on or within 12 months of completing therapy are eligible. Participants with NSCLC and targeted therapy treatment options are eligible for the clinical trial as long as they meet these criteria.

   iv. Participants with recurrent disease > 12 months after adjuvant or neoadjuvant platinum-based chemotherapy, who also subsequently progressed during or after a platinum-doublet regimen and an immune checkpoint inhibitor (given either together or sequentially to treat the recurrence), are eligible v. Participants must have received platinum-based chemotherapy for advanced or metastatic disease and immune checkpoint inhibitor either together (in the same line of treatment) or sequentially (two different lines of treatment) and then progressed.

   k. Non small cell lung cancer combination group i. Non-small cell lung cancer (adenocarcinoma and squamous eligible; endocrine, neuroendocrine and small cell tumors are excluded) ii. Participants must have progressed after at least 1 but not more than 2 prior systemic regimens including chemotherapy and immunotherapy. Participants with NSCLC and targeted therapy treatment options, are eligible for the clinical trial as long as they meet these criteria (progression after 1 or 2 prior therapies). Note: Participants with NSCLC harboring mutations amenable to targeted therapy treatment, are eligible if received targeted therapy as single agent or in combination in 1st or 2nd line of treatment; participants not eligible to receive such therapies in 1st or 2nd line are also eligible to participate to the study.

   iii. Participants who have received adjuvant or neoadjuvant platinum-doublet chemotherapy (after surgery and/or radiation therapy) and an immune checkpoint inhibitor and developed recurrent or metastatic disease while on or within 12 months of completing therapy are eligible iv. Participants with recurrent disease > 12 months after adjuvant or neoadjuvant platinum-based chemotherapy, who also subsequently progressed during or after a platinum-doublet regimen and an immune checkpoint inhibitor (given either together or sequentially to treat the recurrence), are eligible v. Participants must not have received prior taxane therapy either as monotherapy or in combination.

   l. Breast cancer monotherapy group i. HR positive HER2 negative

   • Participant has a histologically and/or cytologically documented diagnosis of HR positive HER2 negative metastatic breast cancer (based on the most recently analyzed tissue sample tested by a local laboratory).
   * Participants must have progressed on at least one line of hormone-based therapy (either alone or in combination) and at least one, but not more than two lines of chemotherapy (including cytotoxic, targeted and/or anti-drug conjugate therapies) for metastatic disease.

   ii. HER2 positive

   • Participant has a histologically and/or cytologically documented diagnosis of HER2 positive metastatic breast cancer (based on the most recently analyzed tissue sample tested by a local laboratory).

   • Participant must have progressed on at least two lines of HER2 targeted therapy for metastatic disease.

   iii. Triple negative breast cancer (TNBC)

   • Participant has a histologically and/or cytologically documented diagnosis of TNBC (based on the most recently analyzed tissue sample tested by a local laboratory).
   * Participants must have progressed on at least two lines of cytotoxic chemotherapy (including cytotoxic, anti-drug conjugate, targeted therapies and/or IO) for metastatic disease.

   Key Exclusion Criteria:

   Participants who meet any of the following criteria will be excluded from the study. The criteria below apply to participants enrolling in Phase 1 or Phase 2.

<!-- -->

1. Active malignancy except for the specific cancer under investigation in this study, ie, participant known to have potentially fatal cancer present for which he/she may be (but not necessarily) currently receiving treatment with the following exceptions:

   1. History of second malignancy that has been successfully treated, with no evidence of active cancer for 3 years prior to enrollment;
   2. Surgically cured low-risk tumors, such as early-stage cervical or endometrial cancer, any cancer in situ, or non-melanoma skin cancers; and
   3. Prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen.
2. Symptomatic and/or untreated CNS metastases or leptomeningeal disease or with primary tumor of CNS origin.

   a. Participants with asymptomatic, previously treated CNS metastases are eligible provided they have been clinically stable for at least 4 weeks and have completed RT> 2 weeks prior to treatment. Participants may be on corticosteroids if on a stable dose equivalent to prednisone 10 mg daily or less.
3. Received anticancer treatment with chemotherapy, antibody therapy or other immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, or experimental drugs ≤ 14 days prior (≤ 28 days prior in case of checkpoint inhibitor therapy and other antibody therapies) to the administration of [177Lu]Lu FAP 2286.
4. Received prior radiopharmaceutical therapy (eg, radium 223 223Ra-dichloride, [177Lu]Lu-DOTA-TATE, [177Lu]Lu-prostate-specific membrane antigen (PSMA)-617, actinium 225 [225Ac]Ac PSMA-617, etc.) or prior EBRT to more than 25% of the bone marrow or received any prior EBRT directly to kidney, or received any EBRT within 2 weeks prior to administration of [177Lu]Lu FAP 2286.

   * Prior administration of a radiopharmaceutical unless 10 or more half-lives have elapsed before injection/infusion of [68Ga]Ga-FAP-2286 or [177Lu]Lu FAP 2286.
5. Ongoing adverse effects from anticancer treatment NCI-CTCAE v5.0 (or higher) Grade 1, with the exception for alopecia and vitiligo.

Exclusion criteria 6 and 7 are removed with Protocol Amendment 7. 8. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

1. Clinically significant and/or uncontrolled cardiac disease such as congestive heart failure requiring treatment (New York Heart Association > Class 2), uncontrolled hypertension, clinically significant arrhythmia, or congenital prolonged QT syndrome;
2. Corrected QT interval (Fridericia's formula) > 450 msec for males or > 470 msec for females at Screening; or
3. Acute coronary syndrome or acute myocardial infarction ≤ 6 months prior to administration of [177Lu]Lu FAP 2286.

   9. Active severe urinary incontinence, severe voiding dysfunction, or urinary obstruction requiring an indwelling/condom catheter that, in the judgment of the investigator, could prevent adhering to radiation safety instructions.

   10. Severe chronic or active HIV infection:

a. Participants on effective antiretroviral therapy with undetectable viral load within 6 months prior to the first dose of [177Lu]Lu FAP 2286 are eligible.

Exclusion criteria 11 and 12 are removed with Protocol Amendment 7. 13. Non-study-related minor surgical procedure ≤ 5 days, or major surgical procedure ≤ 21 days, prior to the administration of [177Lu]Lu FAP 2286; in all cases, the participant must be sufficiently recovered and stable before treatment administration.

14. The following are exclusion criteria, as applicable:

a. Female participants of childbearing potential: i. Refusal to use a highly effective method of contraception or to practice true abstinence during treatment and for 6 months following the last dose of investigational product; ii. Pregnant, suspected pregnancy, or breast feeding; iii. Planning on getting pregnant during treatment and for 6 months following the last dose of investigational product.

b. Male participants with female partners of childbearing potential: i. Refusal to use a highly effective method of contraception or to practice true abstinence during treatment and for 6 months following the last dose of investigational product.

c. All male participants: i. Refusal to use condoms during sex. ii. Planning to make semen donations during treatment and for 6 months following the last dose of investigational product.

15. Significant weight loss (> 10% of body weight) within 28 days prior to providing informed consent for this study.

16. Presence of any other condition that may increase the risk associated with study participation or interfere with the interpretation of study results, and, in the opinion of the investigator, would make the participant inappropriate for entry into the study.

17. Inability to complete the needed investigational and standard imaging examinations due to any reason (e.g., severe claustrophobia, inability to lie still for the entire imaging time).

18. Participants with known hypersensitivity to the active agent or excipients. 19. Severe chronic or active infections (including active tuberculosis, HBV, or HCV infection) requiring systemic antibacterial, antifungal or antiviral therapy within 2 weeks before enrollment.

Note: Antiviral therapy is permitted for participants with chronic HBV or HCV infection. Participants receiving antivirals at Screening should have been treated for > 2 weeks before enrollment. Inactive hepatitis B surface antigen (HbsAg) carriers treated and stable hepatitis B participants (HBV DNA < 500 IU/mL or < 2500 copies/mL) can be enrolled. Participants with detectable hepatitis B surface antigen (HbsAg) or detectable HBV DNA should be managed per treatment guidelines. Participants positive for HCV antibody are eligible only if PCR is negative for HCV RNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose-limiting toxicity (DLTs) | From first dose of study drug through at least 6-8 weeks after end of treatment (up to approximately 2 years)
  To evaluate the safety and tolerability of [177Lu]Lu FAP 2286 and determine the RP2D
Phase 1: recommended Phase 2 dose (RP2D) | From first dose of study drug through at least 6-8 weeks after end of treatment (up to approximately 2 years)
  To evaluate the safety and tolerability of [177Lu]Lu FAP 2286 and determine the RP2D
Phase 1: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) of [177Lu]Lu FAP 2286 | From first dose of study drug through at least 6-8 weeks after end of treatment (up to approximately 2 years)
  To evaluate the safety and tolerability of [177Lu]Lu FAP 2286 and determine the RP2D
Phase 2: Objective Response Rate (ORR) | From date of first [177Lu]Lu FAP 2286 treatment until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 59 months
  Objective response is defined as a best confirmed response of CR or PR by RECIST v1.1 as assessed by the investigator. A confirmed CR or PR is a response that is maintained and documented on a subsequent tumor assessment no less than 28 days after the initial response. For Phase 2, ORR defined as the frequency and percentage of participants with a best confirmed response of CR or PR will be analyzed.
Phase 2: Dose-limiting toxicity (DLTs) | Assessed within 4 weeks of first Lu-FAP2286 treatment
  To evaluate the safety and tolerability of [177Lu]Lu FAP 2286 and determine the RP2D in combination with mFOLFIRINOX in PDAC and the RP2D in combination with nab-paclitaxel in NSCLC (Phase 2 dose escalation for combination therapy)
Phase 2: recommended Phase 2 dose (RP2D) | From first dose of study drug through at least 6-8 weeks after end of treatment (up to approximately 2 years)
  To evaluate the safety and tolerability of [177Lu]Lu FAP 2286 and determine the RP2D in combination with mFOLFIRINOX in PDAC and the RP2D in combination with nab-paclitaxel in NSCLC (Phase 2 dose escalation for combination therapy)
Phase 2: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) of [177Lu]Lu FAP 2286 | From first dose of study drug through at least 6-8 weeks after end of treatment (up to approximately 2 years)
  To evaluate the safety and tolerability of [177Lu]Lu FAP 2286 and determine the RP2D in combination with mFOLFIRINOX in PDAC and the RP2D in combination with nab-paclitaxel in NSCLC (Phase 2 dose escalation for combination therapy)

SECONDARY OUTCOMES:
Phase 1: Absorbed dose (Gy) estimated in organs and tumor lesions | From first dose of study drug until disease progression or end of treatment (up to approximately 9 months)
  To measure the radiation dosimetry of [177Lu]Lu FAP 2286
Phase 1: Maximum standardized uptake value (SUVmax) in tumor lesions | Taken within 2 hours after 68Ga-FAP-2286 IV administration
  To determine tumor uptake using [68Ga]Ga FAP 2286
Phase 1: Comparison of SUVmax in tumor lesions | From time of screening FDG PET/CT to 68Ga-FAP-2286 PET/CT (up to approximately 1 month)
  To evaluate tumor uptake of [68Ga]Ga FAP 2286 as compared to FDG
Phase 1: Concentration of [177Lu]Lu FAP 2286 at the end of infusion (Ceoi) | From first dose of study drug to end of Cycle 6 with (each cycle ~ 6 weeks) (Total Time Frame estimated up to approximately 9 months)
  To evaluate the PK of [177Lu]Lu FAP 2286
Phase 1: Cmax of [177Lu]Lu FAP 2286 | From first dose of study drug to end of Cycle 6 with (each cycle ~ 6 weeks) (Total Time Frame estimated up to approximately 9 months)
  To evaluate the PK of [177Lu]Lu FAP 2286
Phase 1: Tmax of [177Lu]Lu FAP 2286 | From first dose of study drug to end of Cycle 6 with (each cycle ~ 6 weeks) (Total Time Frame estimated up to approximately 9 months)
  To evaluate the PK of [177Lu]Lu FAP 2286
Phase 1: Area under the curve (AUC) of [177Lu]Lu FAP 2286 | From first dose of study drug to end of Cycle 6 with (each cycle ~ 6 weeks) (Total Time Frame estimated up to approximately 9 months)
  To evaluate the PK of [177Lu]Lu FAP 2286
Phase 1: Clearance (CL) of [177Lu]Lu FAP 2286 | From first dose of study drug to end of Cycle 6 with (each cycle ~ 6 weeks) (Total Time Frame estimated up to approximately 9 months)
  To evaluate the PK of [177Lu]Lu FAP 2286
Phase 1: Volume of distribution (Vd) of [177Lu]Lu FAP 2286 | From first dose of study drug to end of Cycle 6 with (each cycle ~ 6 weeks) (Total Time Frame estimated up to approximately 9 months)
  To evaluate the PK of [177Lu]Lu FAP 2286
Phase 1: Half-life (T1/2) of [177Lu]Lu FAP 2286 | From first dose of study drug to end of Cycle 6 with (each cycle ~ 6 weeks) (Total Time Frame estimated up to approximately 9 months)
  To evaluate the PK of [177Lu]Lu FAP 2286
Phase 1: Objective Response Rate (ORR) | From date of first [177Lu]Lu FAP 2286 treatment until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 57 months
  Objective response is defined as a best confirmed response of CR or PR by RECIST v1.1 as assessed by the investigator. A confirmed CR or PR is a response that is maintained and documented on a subsequent tumor assessment no less than 28 days after the initial response.
Phase 1: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) of [68Ga]Ga FAP 2286 | Up to approximately 57 months
  To evaluate the safety and tolerability of [68Ga]Ga FAP 2286.
Phase 2 (Dose expansion): Duration of Response (DoR) | From first documented evidence of CR or PR (the response prior to confirmation) until time of documented disease progression or death due to any cause, whichever comes first, assessed up to approximately 83 months
  Duration of Response (DOR) was defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented radiographic progression or death due to any cause as assessed by investigator according to RECIST v1.1.
Phase 2 (Dose expansion): Disease Control Rate (DCR) | From date of first [177Lu]Lu FAP 2286 treatment until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 83 months
  Disease Control Rate (DCR) is defined as the frequency and percentage of participants with stable disease (SD) of at least 12 weeks (2 consecutive scans with Best Overall Response (BOR) of SD) or a best confirmed response of CR or PR.
Phase 2 (Dose expansion): Progression-free survival (PFS) | From date of first [177Lu]Lu FAP 2286 treatment until date of progression or date of death from any cause, whichever come first, assessed up to 83 months
  Progression-free survival (PFS) is defined as the time from the date of randomization to the date of first evidence of radiographic progression or death due to any cause, whichever occurred first.
Phase 2 (Dose expansion): Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) of [177Lu]Lu FAP 2286 at the RP2D | Up to approximately 83 months
  The distribution of adverse events of [177Lu]Lu FAP 2286 at the RP2D for monotherapy, the RP2D in combination with mFOLFIRNOX in PDAC and the RP2D in combination with nab-paclitaxel in NSCLC will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Phase 2: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) of [68Ga]Ga FAP 2286 | Up to approximately 83 months
  The distribution of adverse events for [68Ga]Ga FAP 2286 will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (19):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Hoag Hospital Irvine, Irvine, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Univ of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Melbourne, Victoria
- Novartis Investigative Site, Montreal, Quebec, Canada
- France (4):
  - Novartis Investigator Site, Montpellier, Cedex 5
  - Novartis Investigator Site, Bordeaux
  - Novartis Investigator Site, Clermont-Ferrand
  - Novartis Investigator Site, Vandœuvre-lès-Nancy
- Novartis Investigative Site, Meldola, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Taunk NK, Escorcia FE, Lewis JS, Bodei L. Radiopharmaceuticals for Cancer Diagnosis and Therapy: New Targets, New Therapies-Alpha-Emitters, Novel Targets. Cancer J. 2024 May-Jun 01;30(3):218-223. doi: 10.1097/PPO.0000000000000720. PMID 38753757